CLINICAL TRIAL: NCT06300268
Title: A Prospective, MulticentRe, Pilot Study to Evaluate the Safety and Performance of The AdvaPro Sirolimus Eluting CorOnary Stent System in Coronary ARtery Stenosis in Indian and European Population(RESTORE)
Brief Title: Advapro Coronary Stent System in Coronary Artery Diseased Patients.
Acronym: RESTORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced MedTech Solutions Pvt. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPL/PL/2023/004
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; De Novo Stenosis Lesion; Coronary Stent Implantation
Keywords: AdvaPro Sirolimus Eluting Coronary Stent System; Late lumen loss; Advanced Medtech Solutions; QCA; PTCA
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Pilot Study (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Other): AdvaPro Sirolimus Eluting Coronary Stent System
  Interventions: Device: AdvaPro Sirolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: AdvaPro Sirolimus Eluting Coronary Stent System — Cardiac Stent

SUMMARY:
A Prospective, Multicentre, Pilot Study to Evaluate the Safety and Performance of the AdvaPro Sirolimus Eluting Coronary Stent System in Coronary Artery Stenosis in Indian and European Population.

To evaluate the performance of AdvaPro Sirolimus Eluting Stent follow up indicated by MACE at 9 months.

Of the 120, 40 patients will be assigned to European population and 80 patients will be assigned to Indian population. QCA is applicable for only in sub-strategy participants at baseline and 9 month follow-up visit.

A QCA Analysis will be performed on minimum 48 patients in Indian population only.

Interval(Days) for patients visit at Day 0, Day 30±6, Day 180±8, Day 270±10 and Day 360±14.

DETAILED DESCRIPTION:
A Prospective, Multicentre, Pilot Study to Evaluate the Safety and Performance of the AdvaPro Sirolimus Eluting Coronary Stent System in Coronary Artery Stenosis in Indian and European Population(RESTORE).

A QCA Analysis will be performed on minimum 48 patients in Indian population only at baseline visit and 9 month follow-up.

Interval(Days) for patients visit at Day 0, Day 30±7, Day 180±8, Day 270±10 and Day 360±14.

Sample size distribution:

Of the 120, 40 patients will be assigned to European population and 80 patients will be assigned to Indian population.

Primary Objective:

To evaluate the performance of AdvaPro Sirolimus Eluting Stent follow up indicated by MACE at 9 months.

Secondary Objectives:

To estimate patient safety and performance through incidence of Major Adverse Cardiac Events (MACE) at 30, 180, 360 days and device oriented composite end point (DOCE), patient oriented composite end point (POCE) Stent Thrombosis, Target vessel failure (TVF), Target Vessel related Myocardial Infarction (TV-MI), and individual components of composite end points at 30, 180, 270 and 360 days after use of AdvaPro Sirolimus Eluting Stent.

To estimate device and procedure success at 30, 180, 270 and 360 days after use of AdvaPro Sirolimus Eluting Stent.

To Estimate Definitive parameters of performance of AdvaPro Sirolimus Eluting Stent as defined by Late Lumen Loss and Diameter Stenosis percentage at 270 days of AdvaPro Sirolimus Eluting Stent.

Exploratory objectives: None

Stent is approved for manufacturing and marketing in India.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Gender : All (Males, Females, Transgenders, Non-binary)
* ICF : Patient or legally authorized representative (LAR) agrees to participation by signing the informed consent form.
* Condition - Clinical : Patient with coronary artery disease Eligible for percutaneous coronary intervention (PCI)
* Condition - Angiographic : Patient with coronary artery disease having one or more de novo stenosis lesion in two native coronary artery with a visually estimated diameter stenosis ≥70%
* Condition - Angiographic : Patients with Reference vessel diameter of 2.5 ~ 3.50 mm
* Condition - Angiographic : Patients with lesion length ≤ 36 mm

Exclusion Criteria:

* Ethical : Pregnant and lactating females
* Patients requiring staged procedure
* Condition : Known congestive heart failure (NYHA IV) or left ventricular ejection fraction (LVEF) <30%
* Condition : Patients with known hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, Sirolimus or similar drugs, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media
* Condition : Current medical condition with a life expectancy of less than 12 months
* Condition : Diagnosis: Acute Myocardial Infarction within 72 hours of Planned Index procedure
* Condition : Patient has current unstable arrhythmias
* Procedural : Patients previously treated with PCI or CABG for any coronary artery lesion revascularization
* Procedural : Patients with Chronic Total Occlusion in two or more vessels
* Procedural : Patients with Ostial lesions (within 5.0mm of vessel origin).
* Procedural : Patients with Bifurcation lesions that include a side branch >2.0 mm diameter
* Procedural : Unprotected Left Main Coronary Artery lesion
* Condition : Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated in opinion of the treating cardiologist
* Condition : Patients with Cardiogenic shock, systemic bleeding and coagulation disorders, intracranial bleeding, Renal insufficiency requiring dialysis, Acute or chronic renal function (serum creatinine >2.0mg/dl or 150 µmol/L), peripheral vascular diseases, cancer, etc. and patients who are planning to undergo surgery within 1 year of the index procedure
* Condition : Patients with platelet count <100.000 cells/mm3 or >700.000 cells/mm3 or a WBC <3.000 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint | 1 Year
  MACE (Hierarchical incidence of Cardiovascular Death, Myocardial infarction or Target Vessel Revascularization)

SECONDARY OUTCOMES:
Incidence of DOCE | 30 Days, 180 Days, 270 Days and 360 days
  1. Cardiovascular Death
  2. Myocardial infarction in the territory of Target vessel
  3. Clinically driven target lesion revascularization
Incidence of POCE | 30 Days, 180 Days, 270 Days and 360 days
  1. All cause death
  2. Any Stroke
  3. Any myocardial infarction
  4. Any revascularization
Incidence of MACE | 30 Days, 180 Days and 360 days
  1. Cardiovascular Death
  2. Non-fatal MI
  3. Target Vessel Revascularization
Target vessel failure (TVF) | 30 Days, 180 Days, 270 Days and 360 days
  Target vessel failure (TVF)
Non-Target Vessel related Myocardial Infarction | 30 Days, 180 Days, 270 Days and 360 days
  Non-Target Vessel related Myocardial Infarction
Stent thrombosis | 0-24 hours, 24 hours-30 days and late 30-365 days
  Stent thrombosis as per
  1. Academic Research Consortium [ARC] Evidence definitions - Definite and probable
  2. As per latency - Acute (0-24 hours), Subacute (24 hours-30 days) and late (30-365 days)
Device success | 0 hour, 24 hours, 3 days
  * Residual coronary stenosis less than 20%
  * Normal coronary flow and absence of coronary dissections > C
  * Procedural and absence of PCI complications including periprocedural MI, coronary perforation, urgent CABG or death or revascularization within 3 days of Index procedure
Procedural Success | 24 Hours
  * Residual Stenosis less than 20%
  * Successful reperfusion of Target vessel region with TIMI Flow ≥ 2
Acute Device Success | 24 Hours
  Acute Device Success as defined by Residual Stenosis ≤ 20%

OTHER OUTCOMES:
For QCA Group | 270 Days
  • Late Lumen Loss
For QCA Group | 270 Days
  • Angiographic binary restenosis
For QCA Group | 270 Days
  • In-stent and in-segment minimum lumen diameter (MLD) and % diameter stenosis (DS)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Philippe Garot, Principal Investigator — Hôpital Privé Jacques Cartier, Massy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abizaid A, Kedev S, Kedhi E, Talwar S, Erglis A, Hlinomaz O, Masotti M, Fath-Ordoubadi F, Lemos PA, Milewski K, Botelho R, Costa R, Bangalore S. Randomised comparison of a biodegradable polymer ultra-thin sirolimus-eluting stent versus a durable polymer everolimus-eluting stent in patients with de novo native coronary artery lesions: the meriT-V trial. EuroIntervention. 2018 Dec 7;14(11):e1207-e1214. doi: 10.4244/EIJ-D-18-00762. PMID 30222120
- [Result] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Result] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Result] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Result] Palmerini T, Biondi-Zoccai G, Della Riva D, Mariani A, Genereux P, Branzi A, Stone GW. Stent thrombosis with drug-eluting stents: is the paradigm shifting? J Am Coll Cardiol. 2013 Nov 19;62(21):1915-1921. doi: 10.1016/j.jacc.2013.08.725. Epub 2013 Sep 11. PMID 24036025
- [Result] Bavry AA, Kumbhani DJ, Helton TJ, Borek PP, Mood GR, Bhatt DL. Late thrombosis of drug-eluting stents: a meta-analysis of randomized clinical trials. Am J Med. 2006 Dec;119(12):1056-61. doi: 10.1016/j.amjmed.2006.01.023. PMID 17145250
- [Result] Scott NA. Restenosis following implantation of bare metal coronary stents: pathophysiology and pathways involved in the vascular response to injury. Adv Drug Deliv Rev. 2006 Jun 3;58(3):358-76. doi: 10.1016/j.addr.2006.01.015. Epub 2006 Mar 6. PMID 16733073
- [Result] Price MJ, Cristea E, Sawhney N, Kao JA, Moses JW, Leon MB, Costa RA, Lansky AJ, Teirstein PS. Serial angiographic follow-up of sirolimus-eluting stents for unprotected left main coronary artery revascularization. J Am Coll Cardiol. 2006 Feb 21;47(4):871-7. doi: 10.1016/j.jacc.2005.12.015. Epub 2006 Jan 6. PMID 16487858
- [Result] Williams DO, Abbott JD, Kip KE; DEScover Investigators. Outcomes of 6906 patients undergoing percutaneous coronary intervention in the era of drug-eluting stents: report of the DEScover Registry. Circulation. 2006 Nov 14;114(20):2154-62. doi: 10.1161/CIRCULATIONAHA.106.667915. Epub 2006 Oct 23. PMID 17060386
- [Result] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Result] Morice MC, Colombo A, Meier B, Serruys P, Tamburino C, Guagliumi G, Sousa E, Stoll HP; REALITY Trial Investigators. Sirolimus- vs paclitaxel-eluting stents in de novo coronary artery lesions: the REALITY trial: a randomized controlled trial. JAMA. 2006 Feb 22;295(8):895-904. doi: 10.1001/jama.295.8.895. PMID 16493102
- [Result] Windecker S, Remondino A, Eberli FR, Juni P, Raber L, Wenaweser P, Togni M, Billinger M, Tuller D, Seiler C, Roffi M, Corti R, Sutsch G, Maier W, Luscher T, Hess OM, Egger M, Meier B. Sirolimus-eluting and paclitaxel-eluting stents for coronary revascularization. N Engl J Med. 2005 Aug 18;353(7):653-62. doi: 10.1056/NEJMoa051175. Epub 2005 Aug 16. PMID 16105989
- [Result] Lemos PA, Moulin B, Perin MA, Oliveira LA, Arruda JA, Lima VC, Lima AA, Caramori PR, Medeiros CR, Barbosa MR, Brito FS Jr, Ribeiro EE, Martinez EE; PAINT trial investigators. Randomized evaluation of two drug-eluting stents with identical metallic platform and biodegradable polymer but different agents (paclitaxel or sirolimus) compared against bare stents: 1-year results of the PAINT trial. Catheter Cardiovasc Interv. 2009 Nov 1;74(5):665-73. doi: 10.1002/ccd.22166. PMID 19670303
- [Result] Goy JJ, Stauffer JC, Siegenthaler M, Benoit A, Seydoux C. A prospective randomized comparison between paclitaxel and sirolimus stents in the real world of interventional cardiology: the TAXi trial. J Am Coll Cardiol. 2005 Jan 18;45(2):308-11. doi: 10.1016/j.jacc.2004.10.062. PMID 15653032
- [Result] Mehilli J, Dibra A, Kastrati A, Pache J, Dirschinger J, Schomig A; Intracoronary Drug-Eluting Stenting to Abrogate Restenosis in Small Arteries (ISAR-SMART 3) Study Investigators. Randomized trial of paclitaxel- and sirolimus-eluting stents in small coronary vessels. Eur Heart J. 2006 Feb;27(3):260-6. doi: 10.1093/eurheartj/ehi721. Epub 2006 Jan 9. PMID 16401670
- [Result] Kandzari DE, Leon MB. Overview of pharmacology and clinical trials program with the zotarolimus-eluting endeavor stent. J Interv Cardiol. 2006 Oct;19(5):405-13. doi: 10.1111/j.1540-8183.2006.00184.x. PMID 17020565
- [Result] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Result] Mauri L, Hsieh WH, Massaro JM, Ho KK, D'Agostino R, Cutlip DE. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med. 2007 Mar 8;356(10):1020-9. doi: 10.1056/NEJMoa067731. Epub 2007 Feb 12. PMID 17296821
- [Result] Ong AT, McFadden EP, Regar E, de Jaegere PP, van Domburg RT, Serruys PW. Late angiographic stent thrombosis (LAST) events with drug-eluting stents. J Am Coll Cardiol. 2005 Jun 21;45(12):2088-92. doi: 10.1016/j.jacc.2005.02.086. PMID 15963413
- [Result] Sousa JE, Costa MA, Abizaid A, Abizaid AS, Feres F, Pinto IM, Seixas AC, Staico R, Mattos LA, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Lack of neointimal proliferation after implantation of sirolimus-coated stents in human coronary arteries: a quantitative coronary angiography and three-dimensional intravascular ultrasound study. Circulation. 2001 Jan 16;103(2):192-5. doi: 10.1161/01.cir.103.2.192. PMID 11208675
- [Result] Sousa JE, Costa MA, Abizaid AC, Rensing BJ, Abizaid AS, Tanajura LF, Kozuma K, Van Langenhove G, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Sustained suppression of neointimal proliferation by sirolimus-eluting stents: one-year angiographic and intravascular ultrasound follow-up. Circulation. 2001 Oct 23;104(17):2007-11. doi: 10.1161/hc4201.098056. PMID 11673337
- [Result] Fajadet J, Wijns W, Laarman GJ, Kuck KH, Ormiston J, Munzel T, Popma JJ, Fitzgerald PJ, Bonan R, Kuntz RE; ENDEAVOR II Investigators. Randomized, double-blind, multicenter study of the Endeavor zotarolimus-eluting phosphorylcholine-encapsulated stent for treatment of native coronary artery lesions: clinical and angiographic results of the ENDEAVOR II trial. Circulation. 2006 Aug 22;114(8):798-806. doi: 10.1161/CIRCULATIONAHA.105.591206. Epub 2006 Aug 14. PMID 16908773
- [Result] Stefanini GG, Byrne RA, Serruys PW, de Waha A, Meier B, Massberg S, Juni P, Schomig A, Windecker S, Kastrati A. Biodegradable polymer drug-eluting stents reduce the risk of stent thrombosis at 4 years in patients undergoing percutaneous coronary intervention: a pooled analysis of individual patient data from the ISAR-TEST 3, ISAR-TEST 4, and LEADERS randomized trials. Eur Heart J. 2012 May;33(10):1214-22. doi: 10.1093/eurheartj/ehs086. Epub 2012 Mar 24. PMID 22447805
- [Result] Dani S, Costa RA, Joshi H, Shah J, Pandya R, Virmani R, Sheiban I, Bhatt S, Abizaid A. First-in-human evaluation of the novel BioMime sirolimus-eluting coronary stent with bioabsorbable polymer for the treatment of single de novo lesions located in native coronary vessels - results from the meriT-1 trial. EuroIntervention. 2013 Aug 22;9(4):493-500. doi: 10.4244/EIJV9I4A79. PMID 23965355
- [Result] Maisel WH. Unanswered questions--drug-eluting stents and the risk of late thrombosis. N Engl J Med. 2007 Mar 8;356(10):981-4. doi: 10.1056/NEJMp068305. Epub 2007 Feb 12. No abstract available. PMID 17296826
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI guideline for percutaneous coronary intervention: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):E266-355. doi: 10.1002/ccd.23390. Epub 2011 Nov 7. No abstract available. PMID 22065485
- [Result] Abizaid A, Costa JR Jr. New drug-eluting stents: an overview on biodegradable and polymer-free next-generation stent systems. Circ Cardiovasc Interv. 2010 Aug;3(4):384-93. doi: 10.1161/CIRCINTERVENTIONS.109.891192. No abstract available. PMID 20716758